CLINICAL TRIAL: NCT07117526
Title: The NUVASCULAR HARBOR Occlusion Device Pilot Study
Brief Title: Nuvascular Harbor Occlusion Device Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuvascular Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-2025-03
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Arterial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: The study population includes adults with intracranial aneurysms (Experimental): Intervention: Aneurysm treatment with the HARBOR Occlusion Device
  Interventions: Device: Aneurysm occlusion with an intrasaccular device

INTERVENTIONS:
Device: Aneurysm occlusion with an intrasaccular device — Intervention with HARBOR Occlusion Device

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the HARBOR Occlusion Device for treating brain aneurysms. The HARBOR Device is investigational (experimental), meaning the Regulatory Authorities have not approved it for commercial use. The data collected in this research study will be used to analyze whether the HARBOR Device is safe and effective in treating brain aneurysms.

DETAILED DESCRIPTION:
Nuvascular is sponsoring a prospective, single-center, single arm clinical trial to assess the safety and effectiveness of the HARBOR Occlusion Device for the treatment of unruptured intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18-79 years of age at the time of screening.
2. Patient must have a single unruptured IA requiring treatment. If the subject has an additional IA requiring treatment, the additional IA must not require treatment within 60 days of the index procedure.
3. The index IA to be treated must have the following characteristics:

   1. Saccular in shape
   2. Diameter 2.5 mm to 12.0 mm
   3. IA is appropriate for treatment with the HARBOR Occlusion Device per device Instructions for Use
4. Patient has an IA that is appropriate for treatment with HARBOR Occlusion Device without the use of additional implanted devices
5. Patient must be able to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule. Patient must sign and date an IRB/EC-approved written informed consent prior to initiation of any study procedures.
6. Patient must sign and date an IRB/EC-approved written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

1. Patient has a ruptured IA, defined as a patient with computed tomography (CT), magnetic resonance imaging (MRI), or lumbar puncture (LP) evidence of subarachnoid hemorrhage attributed to the index aneurysm within the last 180 days.
2. Patient has an IA with characteristics unsuitable for endovascular treatment.
3. Microcatheter could not reach patient's index aneurysm to allow necessary access to treat with study device.
4. Patient has vessel characteristics, tortuosity or morphology which could preclude safe access and support during treatment with study device;
5. Patient has vascular disease or other vascular anomaly so as to preclude the necessary access to the aneurysm for use of the study device.
6. Patient has clinical, angiographic or CT evidence of vasospasm, vasculitis, or intracranial tumor (except small meningioma) or any other intracranial vascular malformations on presentation.
7. Patient has conditions placing them at high risk for ischemic stroke or has exhibited ischemic symptoms such as transient ischemic attacks, minor strokes, or stroke-in-evolution within the prior 60 days.
8. Patient has any circulatory, neurovascular, cardiovascular, or neurologic conditions that have resulted in unstable neurological symptoms.
9. Patient has mRS ≥ 2 prior to presentation
10. Patient has had an SAH from a non-index IA or any other intracranial hemorrhage within 180 days.
11. Patient has physical, neurologic or psychiatric conditions which preclude his/her ability to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule.
12. Patient has a known blood dyscrasia, coagulopathy, or hemoglobinopathy.
13. Patient is pregnant.
14. Patient has known hypersensitivity, which cannot be medically treated, to any component of the study implant device (primarily nickel-titanium alloy), procedural materials, or medications commonly used during the procedure.
15. Patient is concurrently involved in another investigational study or a post-market study that could affect the safety and effectiveness of IA treatment with the study device or with the study's follow-up schedule.
16. Patient has an acute life-threatening illness other than the neurological disease to be treated in this trial.
17. Patient has a life expectancy of less than 2 years due to other illness or condition (in addition to an intracranial aneurysm).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Participants meeting the primary safety and effectiveness endpoints | 10-14 months
  The study's primary effectiveness endpoint is the proportion of subjects with complete aneurysm occlusion without retreatment, recurrent subarachnoid hemorrhage, without significant parent artery stenosis (>50% stenosis) at one year after treatment. A subject will be considered an effectiveness success upon meeting all the above criteria.
  The study's primary safety endpoint is the proportion of subjects with death of any nonaccidental cause or any major stroke (defined as an ischemic or hemorrhagic stroke resulting in an increase of 4 points or more on the National Institutes of Health Stroke Scale) within the first 30 days after treatment or major ipsilateral stroke or death due to neurologic cause from day 31 to the 1 year after treatment. A subject will be considered a safety failure upon meeting any of the above criteria. All safety events will be adjudicated by an independent clinical events committee.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital St. Ivan Rilski, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No